CLINICAL TRIAL: NCT03659565
Title: Increasing Caregiver and Patient Engagement Through an Optimized Personal Health Record
Brief Title: Increasing Caregiver and Patient Engagement Through PHR Use
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual due to Covid-19 restrictions
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0491-18-EP
Record Dates: First submitted 2018-08-01; First posted 2018-09-06 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Pre-Visit Consultation (Experimental): Patients and caregivers will participate in an enhanced pre-visit consultation using Zoom for remote video and audio conferencing with screen sharing capabilities.
  Interventions: Behavioral: Enhanced Pre-Visit Consultation
- Usual Care Control (Active Comparator): Patients continue to receive usual care from their cardiologist.
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: Enhanced Pre-Visit Consultation — The Intervention Group will be given access to the optimized personal health record and will use Zoom as part of the pre-visit consultation.
  Arms: Enhanced Pre-Visit Consultation
Behavioral: Usual Care Control — Caregivers and patients will participate in usual pre-visit process.
  Arms: Usual Care Control

SUMMARY:
Informal caregivers play an integral role in managing complex, chronic disease patients providing services equivalent to an estimated economic value of $470 billion. The inclusion of informal caregivers in the healthcare team can improve care coordination and make health care safer by reducing potential medical errors caused by miscommunication. the investigators reason that a properly designed PHR with a simplified user interface and easy access to relevant content can improve the management of chronic diseases and better integrate caregivers and patients into the healthcare team.

DETAILED DESCRIPTION:
Informal caregivers (caregivers, often family or friends) play an integral role in managing patients with complex, chronic diseases. It is estimated that caregivers provide $470 billion of uncompensated care. Despite their impact, healthcare systems largely neglect caregivers. Long distance caregivers of older adults (who make up 15% of caregivers in America) are at a particular disadvantage. In the current healthcare system, health information technology (HIT) has not been optimized to support the needs of caregivers and patients. Providing HIT that supports enhanced communication between patients, caregivers, and clinicians can improve patient safety by increasing the accuracy of patient data and by reducing miscommunication(1).

There is limited knowledge concerning best practices to promote caregivers' and patients' activation and engagement, especially with HIT. Access to personal health information through the personal health record (PHR) has the potential to improve chronic health care management, and encourage patient engagement. Although caregivers and patients express a willingness to adopt PHRs, in practice, multiple barriers hinder PHR adoption. A properly designed PHR can help caregivers and patients manage their health and become partners in the healthcare team.

This study's overall objective is to identify caregivers and cardiovascular patients' communication and technology needs and to build and test an optimized PHR design that promotes active participation of patients and their caregivers in their health. The overall hypothesis is that an optimized PHR will expand the role of caregivers to improve the patient's health and improve the satisfaction of both patients and caregivers with their care. The investigators will employ an agile, user-centered design process involving caregivers and older cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be patients with heart disease, able read, write, and speak English, and at least 65 years of age.
* Eligible caregivers will be a primary caregiver of an eligible patient, able to read, write, and speak English, and at least 18 years of age.

Exclusion Criteria:

* Individuals under the age of 19 will not be considered for participation.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Patient activation | 12 months
  Patient activation will be measured using Altarum Consumer Engagement (ACE) Measure™. The ACE survey is a 21-item survey that measures patient engagement and health consumerism.
Caregiver activation | 12 months
  Caregiver activation will be measured using the Family Caregiver Activation in Transitions (FCAT) Tool. FCAT is a 10-item tool used to measure caregivers' activation and self-efficacy.

SECONDARY OUTCOMES:
Medication adherence | 12 months
  Medication adherence will be measured using the Medication Adherence Survey (MAS)
Caregiver Satisfaction | 12 months
  Child Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) will be used to measure caregiver satisfaction. HCAHPS is a 62-item survey used to measure that will be modified to measure caregiver satisfaction.
Patient Satisfaction | 12 months
  Consumer Assessment for Healthcare Providers and Systems Survey (CAHPS) will be used to measure patient satisfaction. CAHPS is a 77-item survey used to assess patients' experiences with care.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Clarke, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No